CLINICAL TRIAL: NCT02179658
Title: OPT-80 Phase III Study -A Multi-center, Double Blinded, Randomized, Parallel Group Study To Compare The Safety, Pharmacokinetics And Efficacy of OPT-80 With Vancomycin In Subjects With Clostridium Difficile-Associated Diarrhea (CDAD)
Brief Title: A Study to Compare Safety and Efficacy of OPT-80(Fidaxomicin) With Vancomycin in Subjects With Clostridium Difficile-associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2819-CL-3002
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Clostridium Difficile
Keywords: Clostridium; Infections; Difficile; Vancomycin; Fidaxomicin
MeSH Terms: conditions — Infections | interventions — OPT 80; Fidaxomicin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPT-80 group (Experimental): Oral
  Interventions: Drug: OPT-80
- Vancomycin group (Active Comparator): Oral
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: OPT-80 — oral
  Other Names: fidaxomicin
  Arms: OPT-80 group
Drug: vancomycin — oral
  Arms: Vancomycin group

SUMMARY:
The primary objective of this study is to investigate the safety and efficacy of OPT-80 versus vancomycin in subjects with Clostridium difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, parallel group study. The subjects who meet all of the inclusion criteria and none of the exclusion criteria will be randomized, and will orally receive either OPT-80 twice daily or vancomycin powder four times daily for 10 days. A follow-up investigation will be performed 28 (±3) days after the completion of study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients who have symptoms of CDAD as defined by;

  * (1)Diarrhea: with ≥4 unformed bowel movements (or ≥200 mL unformed stool for subjects having rectal collection devices) and
  * (2)Presence of either toxin A and/or B of C. difficile in the stool
* Subjects who have not received antibacterials (vancomycin, metronidazole, et.al.) aiming at CDAD treatment before the study

Exclusion Criteria:

* Life-threatening or fulminant CDAD
* Ileus paralytic or toxic megacolon
* Likelihood of death before the completion of study from any cause
* Concurrent use of oral vancomycin, metronidazole, et.al. aiming at the treatment of CDAD
* The anticipated need to continue other antibacterials for a period exceeding seven days from providing the informed consent
* Subjects who in the opinion of the investigator require other drugs to control diarrhea
* Need of change in dosage regimen of opiates during the study period
* Need of change in dosage regimen of probiotic products during the study period
* History/complications of ulcerative colitis or Crohn's disease
* Multiple occurrences of CDAD within the past three months
* Hypersensitivity to vancomycin
* Previous exposure to OPT-80 (fidaxomicin)
* Female patients who are pregnant, breastfeeding or possibly pregnant, or wishing to become pregnant during the course of study
* Participation in other clinical research studies or Post Marketing Clinical Trials utilizing an investigational agent within one month prior to providing the informed consent or within five half-lives of the investigational agent, whichever is longer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Global cure rate | Up to 38 days
  Global cure rate is the rate of the subjects satisfying both of the following: being cured at the completion of study drug administration; without recurrence during the follow-up period

SECONDARY OUTCOMES:
Cure rate | Day 10 -11 of the study period
Recurrence rate of CDAD | during the 4-week follow-up period, up to Day 38
Time to resolution of diarrhea | up to 38 days
Microbiological efficacy | Up to 38 days
Plasma concentration of OPT-80(fidaxomicin) | Before administration, Day 1 and Day 10-11
Plasma concentration of OP-1118 | Before administration, Day 1 and Day 10-11
Fecal concentration of OPT-80(fidaxomicin) | Day 10-11
Fecal concentration of OP-1118 | Day 10-11
Safety assessed by the incidence of adverse events, vital signs, ECGs and laboratory tests | Up to 38 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kanto
  - Kinnki
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Mikamo H, Tateda K, Yanagihara K, Kusachi S, Takesue Y, Miki T, Oizumi Y, Gamo K, Hashimoto A, Toyoshima J, Kato K. Efficacy and safety of fidaxomicin for the treatment of Clostridioides (Clostridium) difficile infection in a randomized, double-blind, comparative Phase III study in Japan. J Infect Chemother. 2018 Sep;24(9):744-752. doi: 10.1016/j.jiac.2018.05.010. Epub 2018 Jun 19. PMID 29934056
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=226